CLINICAL TRIAL: NCT02585947
Title: A Multicenter Study to Compare the Efficacy of a Prophylactic Use of Tenofovir by Duration for the Non-Hodgkin's Lymphoma Patients With Isolated Anti-HBc-positivity Who Will be Treated With Rituximab Based Chemotherapy
Brief Title: To Compare the Efficacy of a Prophylactic Use of Tenofovir by Duration for the Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gilead Sciences (Industry); Konkuk University Hospital (Other)
Responsible Party: Principal Investigator, Yoon Jun Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TenoCore
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Non-Hodgkin's Lymphoma, Burkitt's
Keywords: Non-Hodgkin's Lymphoma; Tenofovir
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Non-Hodgkin | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tenofovir for 24 weeks (Experimental): * prophylactic (preemptive) treatment
  * 300mg for 24 weeks
  * once daily
  Interventions: Drug: Tenofovir
- tenofovir for 48 weeks (Experimental): * prophylactic (preemptive) treatment
  * 300mg for 48 weeks
  * once daily
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — Anti-HBc positive patients with Non-Hodgkin's lymphoma planned to receive rituximab based chemotherapy will be randomized to either Group A or Group B in a 1:1 ratio and will be monitored every 12 weeks from the start of treatment for up to 72 weeks after the end of chemotherapy (EOC).
  Other Names: Viread

SUMMARY:
The objective of this study is to analyze factors affecting Hepatitis B Virus (HBV) reactivation in anti-HBc positive patients with Non-Hodgkin's lymphoma treated with rituximab and compare HBV reactivation rates by duration of prophylactic treatment with tenofovir to contribute to the establishment of an effective prevention strategy.

DETAILED DESCRIPTION:
This study will be conducted in a randomized, open-label, multi-center design. On Day 1 of chemotherapy, approximately 90 subjects screened and determined eligible will be randomized to either Group A or Group B in a 1:1 manner for study participation.

* Group A: Upon the EOC, subjects will receive tenofovir 300mg for approximately 6 months (24 weeks) and undergo treatment and follow-up every 12 weeks for up to 72 weeks post chemotherapy.
* Group A: Upon the EOC, subjects will receive tenofovir 300mg for approximately 12 months (48 weeks) and undergo treatment and follow-up every 12 weeks for up to 72 weeks post chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 (Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study during screening to rule out pregnancy. / A woman of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of tenofovir. / If the Investigator obtains information concerning the pregnancy of a female patient, the Investigator must terminate the study drug immediately in that patient, and report the information to IRB in the same manner as for SAE reporting)
2. CD 20 positive patients with Non-Hodgkin's lymphoma who are planned to receive anticancer treatment with rituximab based chemotherapy and A. ECOG performance status 0-2 B. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L) C. Adequate hematological function: hemoglobin ≥ 9g/dL, absolute neutrophil count (ANC) ≥ 1,500/μL, platelet count ≥ 75,000/μL, unless abnormalities are due to bone marrow involvement by lymphoma D. Expected residual life ≥ 6 months
3. Serum HBsAg negative, anti-HCV negative, but anti-HBc positive
4. ALT < 80IU/mL, serum bilirubin < 3.0mg/dL, unless abnormalities are due to liver involvement by lymphoma or tumor lysis syndrome
5. Individuals who were given and understood detailed explanations about this study, voluntarily decided to participate in the study, and provided written informed consent

Exclusion Criteria:

1. Child-Pugh class C
2. Other chronic liver diseases such as autoimmune hepatitis or Wilson's disease
3. Patient who has hypersensitivity to study drug
4. Patient who has galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
5. Patient who is pregnant or on lactating. Or who has plans for pregnant or lactation during study period even the partner of the male patient

Ages: 19 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
HBV reactivation: defined as an increase in HBV DNA at least 10 folds from nadir or reappearance of HBsA or HBeAg in blood during treatment. | after 48 week from the End of treatment

SECONDARY OUTCOMES:
Hepatitis flare: defined as elevation of HBV viral load more than 2,000IU/ml from the baseline or by the reappearance of HBsAg and elevation of ALT at least 100IU/ml from the baseline. | after 48 week from the End of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jang H, Yu SJ, Lee HG, Kim TM, Lee YB, Cho EJ, Lee JH, Yoon JH, Kim YJ. Efficacy of Antiviral Prophylaxis up to 6 or 12 Months From Completion of Rituximab in Resolved Hepatitis B Patients: A Multicenter, Randomized Study. J Korean Med Sci. 2023 Jul 17;38(28):e216. doi: 10.3346/jkms.2023.38.e216. PMID 37463687